CLINICAL TRIAL: NCT01516229
Title: Specific Survey of Norditropin® in Achondroplasia: Survey for Long-term Application
Brief Title: Special Survey for Long Term Application
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-1941
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Achondroplasia
MeSH Terms: conditions — Genetic Diseases, Inborn; Achondroplasia | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Somatropin
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Prescription of somatropin at the discretion of the physician

SUMMARY:
This study is conducted in Japan. The aim of this study is to assess the incidence rate of adverse drug reactions (ADRs) when using somatropin (Norditropin®) for treatment of for achondroplasia without epiphyseal line closure under normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Achondroplasia without epiphyseal line closure

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients being treated with somatropin for achondroplasia without epiphyseal line closure
Sampling Method: Probability Sample
Enrollment: 395 (Actual)
Dates: Start 1997-05-01 (Actual); Primary Completion 2007-03-31 (Actual); Study Completion 2007-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs)

SECONDARY OUTCOMES:
Treatment evaluation using the Foundation for Growth Science's Criteria for Treatment Continuation: Definitely effective, effective, ineffective or definitely ineffective

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com